CLINICAL TRIAL: NCT02200380
Title: A Pilot Study of CDX-301 (rhuFlt3L) With or Without Plerixafor for the Mobilization and Transplantation of Allogeneic Blood Cell Grafts in HLA-Matched Donor/Recipient Sibling Pairs
Brief Title: A Safety and Tolerability Study of CDX-301 With or Without Plerixafor for Stem Cell Mobilization in Matched Related Allogeneic Donor/Recipient Sibling Transplant Pairs
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDX301-03
Record Dates: First submitted 2014-06-16; First posted 2014-07-25 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: For Donors; Related Donors Giving Peripheral Blood Stem Cells (PBSC) to a Sibling; For Recipients; Acute Myelogenous Leukemia (AML); Acute Lymphoblastic Leukemia (ALL); Myelodysplastic Syndrome (MDS); Chronic Myelogenous Leukemia (CML); Non-Hodgkins Lymphoma (NHL); Hodgkins Disease (HD); Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDX-301 (Experimental)
  Interventions: Drug: CDX-301
- CDX-301 and plerixafor (Experimental)
  Interventions: Drug: CDX-301 and plerixafor

INTERVENTIONS:
Drug: CDX-301 — Related donors will receive CDX-301 for 5 days or 7 days.
  Arms: CDX-301
Drug: CDX-301 and plerixafor — Related donors will receive CDX-301 for 5 or 7 days plus plerixafor.
  Arms: CDX-301 and plerixafor

SUMMARY:
This is an open-label, multicenter, prospective pilot study of CDX-301 with or without plerixafor as a stem cell mobilizer for allogeneic transplantation (stem cells that come from another person). HLA-matched sibling healthy volunteers (donors) and patients with protocol specified hematologic malignancies (recipients) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Donors:

* Read, understood and provided written informed consent and willing to comply with all study requirements and procedures
* 6 out of 6 HLA-matched sibling
* Negative test for human immunodeficiency virus (HIV), hepatitis B, and hepatitis C
* Both male and female patients of childbearing potential enrolled in this trial must use adequate birth control measures
* Subjects should be in generally good health and without significant medical conditions, based upon pre-study medical history, physical examination, electrocardiogram (ECG), chest X- ray, and laboratory tests
* Meets all criteria to serve as a mobilized blood cell donor in accordance with all applicable individual Transplant Center criteria

Recipient:

* Read, understood and provided written informed consent and willing to comply with all study requirements and procedures
* 6 out of 6 HLA-matched sibling
* Both male and female patients of childbearing potential enrolled in this trial must use adequate birth control measures

Diagnosis of one of following:

* Acute Myelogenous Leukemia (AML) in 1st remission or beyond
* Acute Lymphoblastic Leukemia (ALL) in 1st remission or beyond
* Chronic Myelogenous Leukemia (CML)
* Chronic Lymphoblastic Leukemia (CLL), relapsing after at least one prior regimen
* Myelodysplastic Syndrome (MDS), either intermediate 1,2, or high risk by IPI Scoring System or transfusion dependent
* Non-Hodgkins Lymphoma (NHL) or Hodgkins Disease (HD) in 2nd or greater complete remission, partial remission, or in relapse
* Meets all criteria to serve as a transplant recipient in accordance with all applicable individual Transplant Center criteria

Exclusion Criteria:

Donors:

* Unwilling or unable to give informed consent, or unable to comply with the protocol including required follow-up and testing
* Prior treatment with any rhuFlt3L product
* Any vaccination within 4 weeks prior to CDX-301 dosing
* Donation of blood within 8 weeks, or donation of plasma within 2 weeks prior to CDX-301 dosing
* Any experimental treatment within 4 weeks prior to CDX-301 dosing
* Use of systemic immunosuppressive agents (excluding topical steroids) within 12 months prior to CDX-301 dosing.
* History of first degree relatives with primary or secondary immunodeficiency to include type 1 diabetes, multiple sclerosis, rheumatoid arthritis, scleroderma or psoriasis
* History of tuberculosis infection
* Herpes zoster within 3 months prior to starting study drug
* Pregnant or nursing

Recipient:

* Unwilling or unable to give informed consent, or unable to comply with the protocol including required follow-up and testing
* Prior allogeneic transplant
* More than one prior autologous transplant
* Prior treatment with any rhuFlt3L product
* Any vaccination within 4 weeks prior to transplant
* Uncontrolled infection at the time of the transplant conditioning regimen
* Pregnant or nursing
* Any condition, which, in the opinion of the clinical investigator, would interfere with the evaluation of the study outcome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-04-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability profile of CDX-301 with or without plerixafor in healthy adult sibling stem cell donors. | 1 Year
  Safety and tolerability will be evaluated by comparing the treatment regimens in regards to vital sign measurements, physical examinations and adverse event reporting.

SECONDARY OUTCOMES:
The proportion of donors whose stem cells can be successfully mobilized and collected with a sufficient CD34+ cell count using CDX-301 with or without plerixafor as the mobilizing agent. | Day 6 - Day 12
  Donor mobilization will be considered successful if ≥ 2 million CD34+ cells/kg recipient weight are collected in no more than two leukapheresis collections.
Describe the cellular composition of allografts mobilized with CDX-301 with or without plerixafor (stem/progenitor cells, T/B/NK-cells). | Day 6 - Day 12
  To describe the cellular composition of allografts mobilized with CDX-301 with or without plerixafor (stem/progenitor cells, T/B/NK-cells).
Incidence of and kinetics of neutrophil and platelet recovery after transplantation of hematopoietic cells mobilized with CDX-301 with or without plerixafor | Day 21, Day 28, Day 56, Day 100, Day 180, Day 270, Day 365.
  To determine the incidence of and kinetics of neutrophil, and platelet recovery after transplantation of hematopoietic cells mobilized with CDX-301 with or without plerixafor.
Incidence of primary and secondary graft failure after transplantation of hematopoietic cells mobilized with CDX301-03 with or without plerixafor. | Day 28, Day 100, Day 180, Day 365.
  To determine the incidence of primary and secondary graft failure after transplantation of hematopoietic cells mobilized with CDX-301 with or without plerixafor.
Rate and quality of immune reconstitution as evidenced by peripheral blood immunophenotype after transplantation of hematopoietic cells mobilized with CDX-301 with or without plerixafor. | Day 28, 100, 180, 365.
  To assess the rate and quality of immune reconstitution as evidenced by peripheral blood immunophenotype after transplantation of hematopoietic cells mobilized with CDX-301 with or without plerixafor.
Incidence of acute and chronic graft-versus host disease (GVHD) after transplantation of hematopoietic cells mobilized with CDX-301 with or without plerixafor. | Day 28, Day 56, Day 100, Day 180, Day 270, Day 365.
  To determine the incidence of acute and chronic graft-versus host disease (GVHD) after transplantation of hematopoietic cells mobilized with CDX-301 with or without plerixafor.
Incidence of CMV reactivation after transplantation of hematopoietic cells mobilized with CDX-301 with or without plerixafor in transplant recipients. | Day 28, Day 56, Day 100, Day 180, Day 270, Day 365.
  To determine the incidence of CMV reactivation after transplantation of hematopoietic cells mobilized with CDX-301 with or without plerixafor in transplant recipients.
Number of post-transplant days of hospitalization in patients that received hematopoietic cells mobilized with CDX-301 with or without plerixafor. | Day 21, 28, 56, 100, 180, 270, 365
  To determine the number of post transplant days of hospitalization after receiving hematopoietic cells mobilized with CDX-301 with or without plerixafor.
Incidence of treatment-related mortality and disease relapse/progression after transplantation of hematopoietic cells mobilized with CDX-301 with or without plerixafor. | Day 21, 28, 56, 100, 180, 270, 365.
  To determine the incidence of treatment-related mortality and disease relapse/progression after transplantation of hematopoietic cells mobilized with CDX-301 with or without plerixafor.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UCLA Medical Center, Los Angeles, California
  - Emory University-Winship Cancer Institute, Atlanta, Georgia
  - Indiana Blood and Marrow Transplant, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Ohio State University Arthur G. James Cancer Hospital and Richard J. Solove Research Institute, Columbus, Ohio
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia